CLINICAL TRIAL: NCT01455480
Title: Trial To Evaluate RPh201 In Treatment Of Partial Thickness Burn
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regenera Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGN-BWH-001
Record Dates: First submitted 2011-10-16; First posted 2011-10-20 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Second Degree Burn Less Than 5%TBSA; Partial Thickness Burn
Keywords: Second Degree Burn; partial thickness burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RPh201 (Experimental)
  Interventions: Drug: RPh201, botanical drug product

INTERVENTIONS:
Drug: RPh201, botanical drug product — topical

SUMMARY:
The objective of this Trial is to evaluate the performance of RPh201 as a treatment for the healing of partial thickness burns. It is further postulated that deep second degree lesions will benefit from the RPh201 treatment promoting granulation and epithelialization as well as wound closure.

DETAILED DESCRIPTION:
The objective of this Trial is to evaluate the performance of RPh201 in the treatment of partial thickness burns (second degree superficial and deep) of less than 5%TBSA.

The additional follow up for a period of 20 weeks will be scheduled to extend the evaluation of wounds of Subjects that completed up to 3 weeks of treatment

This is to include:

* Efficacy assessment of burn improvement following the use of RPh2O1 oil solution administered topically three times per week during an overall treatment period of up to 3 weeks and at the follow-up visit at 20 weeks after end of treatment in Subjects with partial thickness burns (second degree superficial and deep) of less than 5%TBSA
* Safety evaluation of RPh201 formulated as an oil solution administered topically three times per week during an overall treatment period of up to 3 weeks in Subjects with partial thickness burns (second degree superficial and deep) of less than 5%TBSA.

ELIGIBILITY:
Inclusion Criteria:

1. The Subject is 18 years of age and older.
2. The Subject has at least one burn wound or more from 1%- 5% TBSA overall.
3. Subjects defined as a partial thickness burn for conservative treatment (second degree superficial and deep).
4. Subjects will be eligible to participate in the Trial if their target lesion area of the edges is not more than 500-750 cm2 at baseline.
5. The Subject is expected to be available for the 3 weeks Trial ambulatory treatment.
6. The Subject is willing and able to adhere to the protocol regimen.
7. The Subject is able to read, understand, and has signed the informed consent form.

Exclusion Criteria:

1. Electrical and chemical burns wounds that are third degree or full thickness.
2. Burn wounds of more than 48hours from burn event
3. Presence of a systemic infection or significant local infection such as cellulites, purulent drainage, gangrene, or necrosis at the target wound site, as well as nonviable tissue, sinus tracts or tunnels that cannot be removed by debridement.
4. Previous history of any illness or condition that may impair wound healing, immune deficiency or connective tissue disease (e.g., SLE, AIDS), neurological disease (e.g., multiple sclerosis), dialysis due to renal disease and active hepatic disease.
5. Known history for allergy to cottonseed oil or mastic gum
6. Subject is receiving, or has received within one month prior to Visit 1 any treatment known to impair wound healing, including but not limited to: corticosteroids, immuno-suppressive drugs, cytotoxic agents, radiation therapy and chemotherapy.
7. Presence or suspicion of any malignancy.
8. Female Subjects who are pregnant or nursing, or of childbearing potential and are not using adequate contraception.
9. Participation in another clinical trial within 30 days prior to the Screening Visit or during this Trial.
10. Mentally disable Subjects
11. A tourist or foreigner or refugee that cannot be followed for the Trial period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
determine the safety use of RPh201 administered topically three times a week during an overall treatment period of up to 3 weeks | 6 month
  Safety evaluation - To demonstrate safety of using RPh201 oil solution in terms of type and severity of adverse events Achievement of wound closure / epithelialization of more than 75% percent of wound area in up to 3 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Winkler, Dr. MD, Principal Investigator — Clinic of the The Burn Unit, The Department of Plastic & Reconstructive Surgery and Medical Research Infrastructure Development and Health Services Fund by Chaim Sheba Medical Center Tel Hashomer, Israel
Locations (1):
- Clinic of the The Burn Unit, The Department of Plastic & Reconstructive Surgery and Medical Research Infrastructure Development and Health Services Fund by Chaim Sheba Medical Center, Tel Litwinsky, Israel